CLINICAL TRIAL: NCT06703281
Title: Comparison of the Effects of Interscalene Block and Superior Trunk Block on Pulmonary Functions for Shoulder Arthroscopic Surgery Patients
Brief Title: Comparison of the Effects of Interscalene Block and Superior Trunk Block on Pulmonary Functions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Beyza Büyükgebiz Yeşil, MD, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 262d4590-e298-4dfe
Record Dates: First submitted 2024-11-21; First posted 2024-11-25 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Regional Anesthesia Morbidity; Complication Following Peripheral Nerve Block; Phrenic Nerve Paralysis
Keywords: Ultrasound-Guided Nerve or Plane Block; Phrenic Nerve Sparing; Brachial Plexus Block
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The investigator who measures the diaphragmatic excursions and spirometric parameters would be blind to the block type performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interscalene brachial plexus block (Experimental): Patients who underwent shoulder arthroscopic surgery and recieved interscalene brachial plexus block for anesthesia before surgery
  Interventions: Procedure: Interscalene Nerve Block
- Superior trunk brachial plexus block (Experimental): Patients who underwent shoulder arthroscopic surgery and recieved superior trunk brachial plexus block for anesthesia before surgery
  Interventions: Procedure: Superior trunk block

INTERVENTIONS:
Procedure: Interscalene Nerve Block — Patients assigned to the Interscalene Nerve Block would have spirometry and ultrasound-guided diaphragm excursion measurements both pre and post-blok 30 minutes.
  Other Names: Spirometry; Ultrasound
  Arms: Interscalene brachial plexus block
Procedure: Superior trunk block — Patients assigned to the Superior Trunk Nerve Block would have spirometry and ultrasound-guided diaphragm excursion measurements both pre and post-blok 30 minutes.
  Other Names: spirometry; ultrasound
  Arms: Superior trunk brachial plexus block

SUMMARY:
The interscalene block (ISB) is one of the peripheral nerve blocks providing surgical anesthesia and postoperative analgesia in shoulder arthroscopy, eliminating the need for general anesthesia. It is performed by administering local anesthetics (LA) to the C5-C6 roots between the scalene muscles at the level of the cricoid cartilage. ISB-related side effects, such as diaphragmatic paralysis, can occur with the spread of LA to the phrenic nerve over the anterior scalene muscle. To prevent this, a superior trunk block (STB) can be performed by administering LA close to the supraclavicular region where the C5-C6 roots merge into the superior trunk (further away from the phrenic nerve). Although there are studies in the literature demonstrating diaphragmatic paralysis using ultrasound and/or spirometry, no study evaluating diaphragmatic paralysis simultaneously with both ultrasound and spirometry under regional anesthesia alone has been found. Therefore, in this study, the investigators aim to assess the effects of this side effect on diaphragmatic excursion using ultrasound simultaneously and on respiratory functions using spirometry.

DETAILED DESCRIPTION:
Due to diaphragmatic paralysis, interscalene block (ISB) application is contraindicated in patients with pulmonary issues, leaving general anesthesia as the only option. However, the use of opioids for postoperative analgesia in such patients brings unwanted opioid side effects. Consequently, new approaches have emerged to prevent diaphragmatic paralysis, making peripheral blocks feasible for shoulder arthroscopies in patients with pulmonary problems. This study aims to reassess the hypothesis regarding ISB and superior trunk block (STB), routinely used for shoulder arthroscopy surgery, in patients without pulmonary issues, supported by simultaneous ultrasound measurements of diaphragmatic excursion and spirometry measurements of respiratory function. Additionally, the demographic characteristics of patients, onset time of block effects, postoperative additional analgesic requirements, durations of block effects, and times of initial analgesic needs will be observed and compared.

Research Type Description: The study is prospective randomized research. Respiratory function measurements will be taken from patients undergoing ISB and STB, which are routinely performed in brachial plexus blocks in our clinic. These measurements do not involve any invasive procedures and will be solely quantitatively assessed using ultrasound and respiratory function tests.

Case Report Form: The form that will be used is a case report form. Each participant will be assigned a unique number, and all sections related to the study will be completed for each participant.

Data Collection:

After obtaining consent from patients agreeing to participate in the study, patients will be monitored (blood pressure, heart rate, oxygen saturation), and intravenous access will be established.

Dr. Beyza Mehri Büyükgebiz Yeşil will measure diaphragmatic excursion under ultrasound guidance during deep and normal respiration on the side where the block will be performed and record the values in the case report form.

Dr. Beyza Mehri Büyükgebiz Yeşil will perform respiratory function testing with a spirometer and record the values in the case report form.

The blocks will be administered by Assoc Prof Dr. Gökçen Emmez and Prof Dr. İrfan Güngör.

Thirty minutes after the end of the block application, Dr. Beyza Mehri Büyükgebiz Yeşil will measure diaphragmatic excursion under ultrasound guidance during deep and normal respiration on the side where the block was performed and perform respiratory function testing with a spirometer and record the values in the case report form.

Blinding of the study will be ensured by having different researchers perform the block and measurements.

Prof Ulunay Kanatlı will perform the surgical procedure. Patients will be prescribed 3X1 grams of Paracetamol for routine postoperative analgesia.

The onset time of the block effect, postoperative additional analgesic requirements, duration of block effects, and time of initial analgesic needs will be observed and recorded in the case report form.

Both surgeon and patient satisfaction will be recorded in the case report form at the end of surgery. Patients will be contacted by phone one week after discharge to inquire about their current condition.

Data Analysis:

At the end of the study, data will be evaluated via case report forms and interpreted using appropriate statistical methods.

Diaphragmatic excursion change rates will be interpreted and analyzed by Prof. Dr. İrfan Güngör and Prof. Dr. Berrin Günaydın, and respiratory function values from the spirometer will be interpreted and analyzed by Prof. Dr. İpek Kıvılcım Oğuzülgen.

If continuous variables follow a normal distribution, the Student's T-test will be applied; if they do not follow a normal distribution, the Mann-Whitney U test will be applied. The Chi-square test will be applied to compare ratios. Depending on whether the data follows a normal distribution or not, Spearman or Pearson correlation tests will be applied for correlation evaluation. A p value of less than 0.05 will be considered statistically significant. Data will be presented as mean ± standard deviation, median, and n.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective shoulder arthroscopic surgery.
* Age between 18 and 80 years.
* American Society of Anesthesiologists (ASA) physical status I-III.
* Written informed consent obtained.

Exclusion Criteria:

* Refusal to undergo peripheral nerve block.
* Pre-existing peripheral nerve disorders.
* Known respiratory, hepatic, renal, or cardiovascular diseases.
* Allergy to local anesthetics.
* Active infection at the block site.
* Body mass index (BMI) > 40 kg/m².
* Coagulopathy or current anticoagulant therapy.
* Sepsis or systemic infection.
* History of prior surgery at the intended block site.
* Neurological deficits or psychiatric disorders affecting cooperation.
* Inability to perform spirometry or comply with study procedures.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-01-11 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Rate of Hemidiaphragmatic Paralysis | Baseline (pre-block) and 30 minutes post-block.
  Measurement of diaphragmatic excursion (DE) in centimeters using ultrasound during normal and deep breathing. The primary aim is to compare the percentage change in DE between interscalene block (ISB) and superior trunk block (STB) groups. Diagnosis of hemidiaphragmatic paralysis based on diaphragmatic excursion reduction:
  ≥75% reduction classified as complete paralysis, 25-74% reduction as partial paralysis, and
  ≤25% reduction as no paralysis.

SECONDARY OUTCOMES:
Percentage Change in Forced Expiratory Volume in 1 Second (FEV1) and Forced Vital Capacity (FVC) | Baseline (pre-block) and 30 minutes post-block.
  Evaluation of the percentage change in FEV1 and FVC measured with spirometry between ISB and STB groups.
Percentage Change in FEV1/FVC Ratio | Baseline (pre-block) and 30 minutes post-block.
  Evaluation of the percentage change in FEV1/FVC ratio measured with spirometry between ISB and STB groups.
Number of Participants Requiring Additional Analgesics | Intraoperative period and within 24 hours postoperatively.
  Comparison of additional analgesic requirements (e.g., opioids or local anesthetics) between the ISB and STB groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University School of Medicine, Ankara, Turkey (Türkiye)